CLINICAL TRIAL: NCT01636934
Title: A Randomized, Placebo Controlled-Double Blind Study of Minocycline for Reducing the Symptom Burden Produced by Chemoradiation Treatment for Non Small Cell Lung Cancer
Brief Title: Minocycline Study in Non Small Cell Lung Cancer (NSCLC) Patients for Chemoradiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-0347; NCI-2018-01837 (Registry Identifier: NCI CTRP); R01CA026582 (NIH)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non Small Cell Lung Cancer; NSCLC; Symptom Burden; Chemoradiation; CXRT; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn; Placebo; Sugar Pill; Questionnaires; Surveys
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; cyclopia sequence | interventions — Minocycline; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Minocycline (Experimental): Two-arm, placebo-controlled pilot study to obtain preliminary estimates of treatment effects of minocycline in patients with non small cell lung cancer (NSCLC) being consented for concurrent chemoradiation (CXRT). Minocycline 100 mg capsules taken by mouth two times a day every day for 7 weeks, starting on the first week of chemoradiation therapy. Questionnaires at baseline, timepoints during chemoradiation, and at treatment completion for 12 weeks.
  Interventions: Drug: Minocycline; Behavioral: Questionnaires
- Placebo (Placebo Comparator): Two-arm, placebo-controlled pilot study to obtain preliminary estimates of treatment effects of minocycline in patients with non small cell lung cancer (NSCLC) being consented for concurrent chemoradiation (CXRT). Placebo capsules taken by mouth two times a day every day for 7 weeks, starting on the first week of chemoradiation therapy. Questionnaires at baseline, timepoints during chemoradiation, and at treatment completion for 12 weeks.
  Interventions: Other: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Minocycline — 100 mg by mouth two times a day (200 mg/day) every day for 7 weeks, starting on the first week of chemoradiation therapy.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Minocycline
Other: Placebo — 1 capsule by mouth two times a day every day for 7 weeks, starting on the first week of chemoradiation therapy.
  Other Names: sugar pill
  Arms: Placebo
Behavioral: Questionnaires — Questionnaires at baseline, timepoints during chemoradiation, and at treatment completion for 12 weeks.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if minocycline can reduce the side effects reported by patients with NSCLC who are receiving chemoradiation therapy. In this study, minocycline will be compared to a placebo.

Minocycline is an antibiotic that may help to reduce side effects of chemoradiation therapy.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Group 1 will take minocycline. Group 2 will take a placebo.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

You will take the study drug/placebo by mouth, every day during chemoradiation therapy.

You may take the study drug/placebo with a full glass (8 ounces) of water. You may take it with or without food, but if it causes an upset stomach, you should take it with food.

If you have trouble swallowing the dose of study drug/placebo, you can open the capsule right before you take it. You should not lie down for at least 30 minutes after taking the study drug/placebo to reduce the risk of side effects.

You must bring the study drug/placebo container (along with any remaining drug) to every study visit.

Study Visits:

Before you start your chemoradiation treatment:

* You will fill out 4 questionnaires about pain and other symptoms, your tobacco history, your health status, and your quality of life. It should take about 15 minutes to complete all of the questionnaires.
* Blood (about 1 tablespoon) will be drawn for biomarker testing. Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug.

During chemoradiation treatment:

* During Week 1 of chemoradiation, blood (about 1 tablespoon) will be drawn for biomarker testing.
* You will complete the symptom questionnaire in the clinic or by telephone 1 time each week. The symptom questionnaire should take about 5 minutes to complete each time.
* Each week you will be asked about any symptoms you may be having and how they may be affecting your daily activities.

At about Week 4 of chemoradiation:

-You will complete 3 questionnaires about pain and other symptoms, your health status, and your quality of life. It should take about 10 minutes to complete all of the questionnaires.

During the last week of chemoradiation:

* You will complete 4 questionnaires about pain and other symptoms, your health status, your quality of life, and your satisfaction with the study drug/placebo. It should take about 15 minutes to complete all of the questionnaires.
* Blood (about 1 tablespoon) will be drawn for biomarker testing.

After the last week of chemoradiation:

* The study staff will call you 1 time each week to check on you and to complete the pain and symptoms questionnaire at a time that is convenient for you. This phone call should last about 10 minutes. If you have had several side effects from the chemoradiation therapy, this phone call may take longer.
* At about Week 12, blood (about 1 tablespoon) will be drawn for biomarker testing.

End of Study Visit:

Your last study visit will be the same day that you have your last clinic visit with the chemoradiation doctor (around Weeks 12-13). At this visit, you will complete the pain and other symptoms questionnaire, the health status questionnaire, and the smoking questionnaires. It should take about 10 minutes to complete all questionnaires.

Length of Study:

You will be on study for up to 13 weeks. You will take the study drug/placebo every day during chemoradiation treatment, and continue to complete the questionnaires until 12-13 weeks. You will be taken off study early if you have intolerable side effects or the study doctor thinks it is in your best interest.

This is an investigational study. Minocycline is FDA approved and commercially available for the treatment of bacterial infection. Using minocycline to treat side effects of chemoradiation treatment in patients with NSCLC is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologically proven diagnosis of NSCLC and consented to receive CXRT at MD Anderson
2. Patients > or = 18 years old
3. Patients who will receive CXRT with platinum/taxane-based chemotherapy and with a total radiation dose of >or = 50 Gy, per treating physician's assessment
4. Patients who speak English or Spanish (due to MDASI language options, we are only accruing English-speaking or Spanish-speaking patients to the protocol)
5. Patients willing and able to review, understand, and provide written consent before starting therapy
6. Patients with normal renal function according to MD Anderson testing standards and no prior renal disease [screening cut off for serum creatinine < 1.5 times ULN]
7. Patients must have the following screening results for hepatic function according to MD Anderson testing standards: total bilirubin < 1.5 times the upper limit of normal; alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST - if available) must be < 2 times the upper limit of normal

Exclusion Criteria:

1. Patients with a history of clinically significant cutaneous drug reaction to minocycline, as documented in the patient medical records
2. Patients who are enrolled in other symptom management or symptom clinical trials
3. Patients who currently have bile duct obstruction or cholelithiasis
4. Patients with hypersensitivity to any tetracyclines
5. Patients who are pregnant; pregnancy will be confirmed by negative urine test
6. Patients on vitamin K antagonist warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 22, 2013 to August, 19 2015. All recruitment done at the University of Texas MD Anderson Cancer
Pre-assignment Details: Of the 51 participants enrolled 2 participant were excluded from the study before assignment to groups.
Groups:
- Minocycline: Minocycline 100 mg twice a day during standard of care chemoradiation therapy plus additional follow up for 5 weeks, for a total of 12 weeks.
- Placebo: Placebo 100 mg twice a day during during standard of care chemoradiation plus additional follow up for 5 weeks, for a total of 12 weeks.
Period: Overall Study
Arm/Group | Minocycline | Placebo
Started | 25 | 24
Completed | 19 | 21
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Chemo cancel | 1 | 0
Not completed — Too ill to continue | 1 | 0
Not completed — Never started study medication | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 6 | 19
  >=65 years | 6 | 15 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.1) | 67.3 (6.3) | 64.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: AUC Value Symptom Severity Differences
Description: Primary outcome variable for this trial will be the mean difference between AUC values recorded for patients assigned to the treatment and control arms. AUC values calculated for the five M.D. Anderson Symptom Inventory (MDASI) items corresponding to fatigue, pain, disturbed sleep, lack of appetite, and sore throat. AUC is sum of the area of the trapezoids that can be fitted during the 12 week period and is measured in units of mean MDASI score in days. Each item is rated on a 0 to 10 scale with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imagine or complete interference.
Time Frame: up to 12 weeks
Population: Of the 49 randomized patients, 40 were evaluable for the primary efficacy analysis
Measure: Mean (Standard Deviation); unit: Units on a scale *week
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 19 | 21
Units on a scale *week
  Fatigue | 31.18 (14.22) | 44.98 (20.9)
  Pain | 17.13 (12.4) | 26.64 (21.56)
  Disturbed Sleep | 17.34 (14.29) | 19.5 (16.41)
  Lack of Appetite | 17.16 (15.76) | 27.31 (24.95)
  Soar Throat | 4.45 (7.23) | 4.36 (9.51)

2. Secondary Outcome: Number of Participants With Treatment-Induced Inflammatory Response
Description: To examine the effectiveness of minocycline in reducing treatment-induced inflammatory response (serum C-reactive protein (CRP), interleukin (IL)-6, TNF-a, sTNF-R1, sTNF-R2, and activation of indoleamine 2,3-dioxygenase (IDO)).
Time Frame: up to 12 weeks
Population: The blood sample collection was an optional procedure for the participants no data were not collected.
Arm/Group | Minocycline | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of the study medication, up to 30 days after last dose administered.
Arm/Group | Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT01636934/Prot_SAP_000.pdf